CLINICAL TRIAL: NCT05653518
Title: Using Closed-Loop Artificial Pancreas Technology to Reduce Glycemic Variability and Subsequently Improve Cardiovascular Health in Type 1 Diabetes
Brief Title: Artificial Pancreas Technology to Reduce Glycemic Variability and Improve Cardiovascular Health in Type 1 Diabetes
Acronym: WBH002
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, William Horton, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220180; 941481 (Other Grant/Funding Number: American Heart Association); 3-SRA-2023-1236-M-B (Other Grant/Funding Number: Juvenile Diabetes Research Foundation)
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes
Keywords: Glycemic Variability; Inflammation; Oxidative Stress; Endothelial Function; Myocardial Perfusion; Aortic Stiffness; Flow-Mediated Dilation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Inflammation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Closed-loop artificial pancreas (AP) (Experimental): FDA approved Tandem t:slim insulin pump with Control-IQ Technology and the Dexcom G6 CGM
  Interventions: Device: Tandem t:slim X2 with Control-IQ Technology
- Sensor Augmented Pump (SAP) therapy (Experimental): Sensor augmented pump (SAP) therapy that includes the use of a study CGM and the participant's current insulin therapy (i.e., either insulin pump or multiple daily injections)
  Interventions: Device: Sensor augmented pump (SAP) therapy

INTERVENTIONS:
Device: Tandem t:slim X2 with Control-IQ Technology — FDA approved Tandem t:slim insulin pump with Control-IQ Technology and the Dexcom G6 CGM
  Arms: Closed-loop artificial pancreas (AP)
Device: Sensor augmented pump (SAP) therapy — Sensor augmented pump (SAP) therapy that includes the use of a study CGM and the participant's personal insulin pump
  Arms: Sensor Augmented Pump (SAP) therapy

SUMMARY:
This study will examine the potential cardiovascular effect(s) of artificial pancreas (AP) technology in patients with type 1 diabetes. AP technology is a system of devices that closely mimics the glucose-regulating function of a healthy human pancreas. It includes an insulin pump and a continuous glucose monitor (CGM). In this study, the investigators will research whether improvements in blood glucose levels and blood glucose variability will in turn decrease biomarkers of inflammation and endothelial dysfunction while improving cardiovascular function.

DETAILED DESCRIPTION:
Cardiovascular disease is a type of disease that affects the heart and blood vessels. The current care for cardiovascular disease prevention in people with type 1 diabetes is to manage blood pressure, cholesterol blood levels, or manage blood glucose levels.

This study will examine the potential cardiovascular effect(s) of artificial pancreas (AP) technology in patients with type 1 diabetes. AP technology is a system of devices that closely mimics the glucose-regulating function of a healthy human pancreas. It includes an insulin pump and a continuous glucose monitor (CGM). In this study, we will use the Food and Drug Administration (FDA)-approved Tandem t:slim insulin pump with Control-IQ Technology and the FDA approved Dexcom G6 CGM. This study will research whether improvements in blood glucose metrics lead to reductions in some of the cardiovascular biomarkers that represent harmful effects in people with type 1 diabetes. Subjects will be randomly assigned to one of two study groups for 12 weeks---Group 1 will be treated with AP Technology and Group 2 will wear the study CGM and continue to use their current diabetes management strategy (i.e., standard care).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on World Health Organization criteria, of type 1 diabetes for at least one year
2. Currently using insulin for at least six months
3. Ages 18-≤40 years
4. Hemoglobin A1c <10.5%
5. Body mass index 18-30 kg/m2
6. Blood pressure <140/90 mmHg
7. For females, not currently known to be pregnant or breastfeeding
8. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued
9. Both pump and MDI users will use insulin parameters such as carbohydrate ratio and correction factors consistently in order to dose insulin for meals or corrections; pump users will have history of entering this information into their pump
10. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
11. Access to internet and willingness to upload data during the study as needed, including data generated prior to the start of the study
12. Current use of a glucometer that is downloadable; or willingness to use a study glucometer
13. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol
14. Willingness to use personal lispro (Humalog) or aspart (Novolog) and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study
15. Total daily insulin dose (TDD) at least 10 U/day.
16. Willingness not to start any new non-insulin glucose-lowering agent during the trial

Exclusion Criteria:

1. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
2. Diagnosis of diabetic ketoacidosis in the 12 months prior to enrollment
3. Prior diagnosis of cardiac disease (e.g., myocardial infarction, congestive heart failure)
4. Cerebrovascular accident in the 12 months prior to enrollment
5. Uncontrolled resting arterial hypertension
6. Conditions that would make use of a CGM difficult (e.g., blindness, severe arthritis, immobility)
7. Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
8. Concurrent use of any non-insulin glucose-lowering agent (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, and/or sulfonylureas)
9. Hemophilia or any other bleeding disorder
10. Currently being treated for a seizure disorder
11. A medical condition or medication, which in the opinion of the investigator or designee, would put the participant or study at risk
12. Current smokers or those who have quit smoking <2 years ago
13. Screening Electrocardiogram (ECG) findings indicative of arrhythmia, sinus node disease, or ischemic heart disease
14. Any woman with hemoglobin (Hgb) <11 g/dL or any man with Hgb <12 g/dL on screening laboratory evaluation (i.e., complete blood count)
15. History of hypersensitivity or prior adverse reaction (e.g., anaphylaxis or angioedema) to IV regular insulin infusion
16. Diagnosis of peripheral neuropathy (assessed by monofilament examination), macroalbuminuria (urine albumin:creatinine >300 mg per g), or retinopathy beyond mild, nonproliferative retinopathy
17. Unstable (i.e., dose adjustment less than 4 weeks prior to study enrollment) doses of vasoactive medications (e.g., calcium channel blockers, statins, nitrates, alpha-blockers, beta-blockers, ACE inhibitors, etc.)
18. History of hypersensitivity or prior adverse reaction to Definity microbubble infusion
19. Current enrollment in another clinical trial, unless approved by the investigator of both studies or if clinical trial is a non-interventional registry trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Glucose Time-in-Range | 12 weeks
  Time-in-range will measured by continuous glucose monitor device

SECONDARY OUTCOMES:
High-sensitivity C-reactive protein (hs-CRP) | At baseline (0 weeks), 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Inflammatory Biomarker
TNF-alpha | At baseline (0 weeks), 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Inflammatory Biomarker
Interleukin-6 (IL-6) | At baseline (0 weeks), 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Inflammatory Biomarker
E-selectin | At baseline (0 weeks), 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Biomarker of endothelial dysfunction
Intracellular adhesion molecule 1 (ICAM-1) | At baseline (0 weeks), 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Biomarker of endothelial dysfunction
Myocardial Perfusion (measured by contrast-enhanced ultrasound [CEU]) | At baseline and 12 weeks of treatment
  CEU will be assessed before and during a euglycemic-hyperinsulinemic clamp
Carotid Femoral Pulse Wave Velocity (cfPWV) | At baseline and 12 weeks of treatment
  Measurement of change in central aortic stiffness
Brachial artery flow-mediated dilation (FMD) | At baseline and 12 weeks of treatment
  Measure of conduit artery endothelial function
Insulin sensitivity | At baseline and 12 weeks of treatment
  insulin sensitivity will be assessed by M value during a euglycemic-hyperinsulinemic clamp

OTHER OUTCOMES:
Human CD14+CD16- monocytes | At baseline (0 weeks), 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Proinflammatory immune cells associated with atherosclerosis

CONTACTS AND LOCATIONS:
Overall Officials: William B Horton, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Livingstone SJ, Looker HC, Hothersall EJ, Wild SH, Lindsay RS, Chalmers J, Cleland S, Leese GP, McKnight J, Morris AD, Pearson DW, Peden NR, Petrie JR, Philip S, Sattar N, Sullivan F, Colhoun HM. Risk of cardiovascular disease and total mortality in adults with type 1 diabetes: Scottish registry linkage study. PLoS Med. 2012;9(10):e1001321. doi: 10.1371/journal.pmed.1001321. Epub 2012 Oct 2. PMID 23055834
- [Background] Secrest AM, Becker DJ, Kelsey SF, Laporte RE, Orchard TJ. Cause-specific mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes. Diabetes. 2010 Dec;59(12):3216-22. doi: 10.2337/db10-0862. Epub 2010 Aug 25. PMID 20739685
- [Background] Martin-Timon I, Sevillano-Collantes C, Segura-Galindo A, Del Canizo-Gomez FJ. Type 2 diabetes and cardiovascular disease: Have all risk factors the same strength? World J Diabetes. 2014 Aug 15;5(4):444-70. doi: 10.4239/wjd.v5.i4.444. PMID 25126392
- [Background] Priya G, Kalra S. A Review of Insulin Resistance in Type 1 Diabetes: Is There a Place for Adjunctive Metformin? Diabetes Ther. 2018 Feb;9(1):349-361. doi: 10.1007/s13300-017-0333-9. Epub 2017 Nov 14. PMID 29139080
- [Background] Alessa T, Szeto A, Chacra W, Mendez A, Goldberg RB. High HDL-C prevalence is common in type 1 diabetes and increases with age but is lower in Hispanic individuals. J Diabetes Complications. 2015 Jan-Feb;29(1):105-7. doi: 10.1016/j.jdiacomp.2014.08.011. Epub 2014 Sep 6. PMID 25441221
- [Background] Norgaard K, Feldt-Rasmussen B, Borch-Johnsen K, Saelan H, Deckert T. Prevalence of hypertension in type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1990 Jul;33(7):407-10. doi: 10.1007/BF00404089. PMID 2401396
- [Background] Corbin KD, Driscoll KA, Pratley RE, Smith SR, Maahs DM, Mayer-Davis EJ; Advancing Care for Type 1 Diabetes and Obesity Network (ACT1ON). Obesity in Type 1 Diabetes: Pathophysiology, Clinical Impact, and Mechanisms. Endocr Rev. 2018 Oct 1;39(5):629-663. doi: 10.1210/er.2017-00191. PMID 30060120
- [Background] Kanter JE, Shao B, Kramer F, Barnhart S, Shimizu-Albergine M, Vaisar T, Graham MJ, Crooke RM, Manuel CR, Haeusler RA, Mar D, Bomsztyk K, Hokanson JE, Kinney GL, Snell-Bergeon JK, Heinecke JW, Bornfeldt KE. Increased apolipoprotein C3 drives cardiovascular risk in type 1 diabetes. J Clin Invest. 2019 Jul 11;129(10):4165-4179. doi: 10.1172/JCI127308. PMID 31295146
- [Background] Risso A, Mercuri F, Quagliaro L, Damante G, Ceriello A. Intermittent high glucose enhances apoptosis in human umbilical vein endothelial cells in culture. Am J Physiol Endocrinol Metab. 2001 Nov;281(5):E924-30. doi: 10.1152/ajpendo.2001.281.5.E924. PMID 11595647
- [Background] Quagliaro L, Piconi L, Assaloni R, Martinelli L, Motz E, Ceriello A. Intermittent high glucose enhances apoptosis related to oxidative stress in human umbilical vein endothelial cells: the role of protein kinase C and NAD(P)H-oxidase activation. Diabetes. 2003 Nov;52(11):2795-804. doi: 10.2337/diabetes.52.11.2795. PMID 14578299
- [Background] Piconi L, Quagliaro L, Assaloni R, Da Ros R, Maier A, Zuodar G, Ceriello A. Constant and intermittent high glucose enhances endothelial cell apoptosis through mitochondrial superoxide overproduction. Diabetes Metab Res Rev. 2006 May-Jun;22(3):198-203. doi: 10.1002/dmrr.613. PMID 16453381
- [Background] Horvath EM, Benko R, Kiss L, Muranyi M, Pek T, Fekete K, Barany T, Somlai A, Csordas A, Szabo C. Rapid 'glycaemic swings' induce nitrosative stress, activate poly(ADP-ribose) polymerase and impair endothelial function in a rat model of diabetes mellitus. Diabetologia. 2009 May;52(5):952-61. doi: 10.1007/s00125-009-1304-0. Epub 2009 Mar 5. PMID 19263033
- [Background] Frontoni S, Di Bartolo P, Avogaro A, Bosi E, Paolisso G, Ceriello A. Glucose variability: An emerging target for the treatment of diabetes mellitus. Diabetes Res Clin Pract. 2013 Nov;102(2):86-95. doi: 10.1016/j.diabres.2013.09.007. Epub 2013 Sep 25. PMID 24128999
- [Background] Ayano-Takahara S, Ikeda K, Fujimoto S, Hamasaki A, Harashima S, Toyoda K, Fujita Y, Nagashima K, Tanaka D, Inagaki N. Glycemic variability is associated with quality of life and treatment satisfaction in patients with type 1 diabetes. Diabetes Care. 2015 Jan;38(1):e1-2. doi: 10.2337/dc14-1801. No abstract available. PMID 25538320
- [Background] FLAT-SUGAR Trial Investigators. Glucose Variability in a 26-Week Randomized Comparison of Mealtime Treatment With Rapid-Acting Insulin Versus GLP-1 Agonist in Participants With Type 2 Diabetes at High Cardiovascular Risk. Diabetes Care. 2016 Jun;39(6):973-81. doi: 10.2337/dc15-2782. Epub 2016 Apr 19. PMID 27208320
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Brown SA, Kovatchev BP, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, Laffel LM, Levy CJ, Pinsker JE, Wadwa RP, Dassau E, Doyle FJ 3rd, Anderson SM, Church MM, Dadlani V, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Kollman C, Beck RW; iDCL Trial Research Group. Six-Month Randomized, Multicenter Trial of Closed-Loop Control in Type 1 Diabetes. N Engl J Med. 2019 Oct 31;381(18):1707-1717. doi: 10.1056/NEJMoa1907863. Epub 2019 Oct 16. PMID 31618560
- [Background] Hovorka R, Kumareswaran K, Harris J, Allen JM, Elleri D, Xing D, Kollman C, Nodale M, Murphy HR, Dunger DB, Amiel SA, Heller SR, Wilinska ME, Evans ML. Overnight closed loop insulin delivery (artificial pancreas) in adults with type 1 diabetes: crossover randomised controlled studies. BMJ. 2011 Apr 13;342:d1855. doi: 10.1136/bmj.d1855. PMID 21493665
- [Background] Kovatchev B, Anderson SM, Raghinaru D, Kudva YC, Laffel LM, Levy C, Pinsker JE, Wadwa RP, Buckingham B, Doyle FJ 3rd, Brown SA, Church MM, Dadlani V, Dassau E, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Lum J, Beck RW; iDCL Study Group. Randomized Controlled Trial of Mobile Closed-Loop Control. Diabetes Care. 2020 Mar;43(3):607-615. doi: 10.2337/dc19-1310. Epub 2020 Jan 14. PMID 31937608
- [Background] Miller RG, Secrest AM, Sharma RK, Songer TJ, Orchard TJ. Improvements in the life expectancy of type 1 diabetes: the Pittsburgh Epidemiology of Diabetes Complications study cohort. Diabetes. 2012 Nov;61(11):2987-92. doi: 10.2337/db11-1625. Epub 2012 Jul 30. PMID 22851572